CLINICAL TRIAL: NCT02868372
Title: The Efficacy of Swabbing of Subcutaneous Tissues of Cesarean Section Wounds With Povidone Iodine to Prevent Postoperative Wound Infection: A Randomized Controlled Clinical Trial
Brief Title: Swabbing of Subcutaneous Tissues of Cesarean Section Wounds With Povidone Iodine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam Rashad Abdel-Hafeez Othman, Associate professor, OB-GYN department- Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AUH2
Record Dates: First submitted 2016-07-29; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Wound Infection
Keywords: Cesarean section; Betadine; Wound infection
MeSH Terms: conditions — Wound Infection | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betadine group (Active Comparator): Subcutaneous tissues of cesarean section wounds are swabbed with10% undiluted Povidone Iodine solution without mobbing before closure of subcutaneous tissues
  Interventions: Drug: Povidone iodine
- No intervention group (No Intervention): No swabbing of subcutaneous tissue of cesarean section wounds

INTERVENTIONS:
Drug: Povidone iodine — After closure of the anterior wall of the rectus sheath, the subcutaneous tissues of the cesarean section wound will be swabbed with 10% undiluted Povidone iodine without mobbing.
  Other Names: Betadine
  Arms: Betadine group

SUMMARY:
The study has 2 groups. Group A in which the subcutaneous tissue will be swabbed with 10 cc of undiluted 10% povidone iodine and will not be mobbed. Group B ; No swabbing. Women in both groups will be followed up during hospital stay and outpatient clinic visits a week and a month after cesarean delivery for surgical site complications which will be evaluated by the researcher.

DETAILED DESCRIPTION:
Aim of the study:

To assess the efficacy of subcutaneous swabbing of cesarean section wounds with povidone iodine to prevent postoperative wound infection.

Study Design: Randomized controlled trial.

Subjects: Women having a cesarean delivery.

The women will have a full description of the study and Subjects will be randomized by selecting a sequentially numbered sealed envelope to one of each group which will be opened during closure of rectus sheath.

Method :

* Patient will receive single dose of prophylactic antibiotic (2-grams first generation cephalosporin) intravenous at time of cesarean delivery during induction of anesthesia. -The same type of suturing material; vicryl No1 will be used for rectus Sheath repair in both groups.
* The same type of suturing material will be used to suture the subcutaneous tissue and the skin (vicryl NO 2/0).

Follow up : Women in both groups will be followed up during hospital stay and outpatient clinic visits a week and a month after cesarean delivery for surgical site complications which will be evaluated by the researcher.

Outcome :The study outcome is to detect and record the incidence of surgical wound infection in both groups.It is a composite outcome with presence of any of the following is considered infection:

* Induration
* Swelling of the wound edges
* Discharge of pus or wound dehiscence.
* Purulent drainage with or without laboratory confirmation, from the superficial incision
* Pain or tenderness with redness, or heat
* Superficial incision being deliberately opened by surgeon.

Sample size estimation:

It was calculated that 269 patients are required in each arm to detect a 5% reduction (from 7% to 2%) in cesarean section wound infection rates between study and control groups.

Statistical Analysis:

Data will be tabulated using Statistical Package for Social Scientists (SPSS) program and statistical analysis will be carried out with suitable statistical tests. Continuous variables will be presented as mean and standard deviation, and will be compared using Student-t-test. Dichotomous variables will be compared using Chi square and the cut off point for P-value will be less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All women having either first time or repeat cesarean section whether elective or emergency.

Exclusion Criteria:

* Women with prolonged rupture of membranes more than 12 hours.
* Women with morbid obesity with BMI>35.
* Women with diabetes, hypertension or anemia with hemoglobin<9.
* Women on corticosteroid therapy or immunosuppressed women.
* Women with intraoperative hemorrhage or hematoma formation.
* Women allergic to betadine.
* The cesarean section which duration exceed one hour or associated with other surgical procedure.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 538 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Detect and record the incidence of surgical wound infection in both groups | One month
  : Women in both groups will be followed up during hospital stay and outpatient clinic visit for one month after cesarean delivery for surgical site complications which will be evaluated by the researcher

IPD SHARING:
Plan to Share IPD: No